CLINICAL TRIAL: NCT05113563
Title: Investigation of TEST (Transcranial Electric Stimulation Therapy) for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Diana Martinez, Clinical Professor in Psychaitry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 7978
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- open label (Other): this is an open label study
  Interventions: Device: Transcranial Electric Stimulation Therapy

INTERVENTIONS:
Device: Transcranial Electric Stimulation Therapy — TEST is a form of brain stimulation.

SUMMARY:
The goal in this study is to investigate TEST (Transcranial Electric Stimulation Therapy) for chronic pain. It requires an inpatient stay on our research unit of about a month. The study is designed to address the cognitive and emotional aspects of chronic pain and other conditions that often accompany this disorder, such as major depression or drug use.

DETAILED DESCRIPTION:
This project proposes to investigate the feasibility of TEST in subjects with chronic pain. This will be an open-label study where subjects (n=12) are administered 8-10 sessions of TEST over 4 weeks. Measurements of pain, mood, and memory will be obtained before and after the sessions. The hypothesis is that TEST will be feasible and tolerable in this population.

ELIGIBILITY:
Inclusion Criteria:

1. adults (ages 22 to 60) who understand all procedures and have the ability to provide informed consent, with a score on the Mini-Mental Status Exam of at least 24;
2. participants experiencing chronic pain, with ongoing pain symptoms, and score on the Brief Pain Inventory of > 5 on question #3 (which asks about maximal pain in the past 24 hours) or > 5 on question #5 (which asks about average pain in the past 24 hours);
3. a diagnosis of chronic postoperative pain, low back pain, musculoskeletal pain, fibromyalgia, visceral pain or neuropathic pain, including complex regional pain syndrome or peripheral neuropathy;
4. no significant changes in pain medications for at least one month prior to study entry.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Group: All participants received open label TEST
Period: Overall Study
Arm/Group | Active Group
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Group
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 2
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Number enrolled in study who completed [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Will be Assessed by the Percent of Participants Who Complete
Description: Feasibility will be assessed by the percent of participants start study procedures and complete these
Time Frame: 4 weeks
Population: all participants entered to study procedures
Measure: Count of Participants; unit: Participants
Arm/Group | Active Group
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 1 month
Description: Definition was not different from clinical trials.gov
Arm/Group | Active Group
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Group (N=6)
participant experienced symptoms from stopping medication (not a study procedure) (Musculoskeletal and connective tissue disorders) | 1 (1) — The participant abruptly stopped a medications and experience unusual paresthesias. This was not part of the study procedures, occurred during the follow up, and was not study related.
participant experienced fatigue and depressed mood after taking medication (not a study procedure) (Psychiatric disorders) | 1 (1) — During the follow up (after all study interventions completed) a participant attended an appointment with her physician and was prescribed an off label medication. She experienced fatigue and depressed mood from this. The event was not study related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT05113563/Prot_SAP_000.pdf